CLINICAL TRIAL: NCT01994031
Title: Dose Escalation and Pharmacokinetic Study of Paclitaxel Liposome Injection in Treating Patients With Advanced Solid Tumor After Failure From Conventional Treatments
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Luye Sike Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJLYSK-LPS-2013-01
Record Dates: First submitted 2013-10-31; First posted 2013-11-25 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Solid Tumors
Keywords: paclitaxel liposome injection; paclitaxel
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Dose level A (Experimental): Paclitaxel liposome injection 135mg/m2 on day 1, First cycle 28 days and subsequent cycles each 21 days
  Interventions: Drug: Paclitaxel liposome injection
- Dose level B (Experimental): Paclitaxel liposome injection 175mg/m2 on day 1, First cycle 28 days and subsequent cycles each 21 days
  Interventions: Drug: Paclitaxel liposome injection
- Dose level C (Experimental): Paclitaxel liposome injection 210mg/m2 on day 1, First cycle 28 days and subsequent cycles each 21 days
  Interventions: Drug: Paclitaxel liposome injection
- Dose level D (Experimental): Paclitaxel liposome injection 250mg/m2 on day 1, First cycle 28 days and subsequent cycles each 21 days
  Interventions: Drug: Paclitaxel liposome injection
- Dose level E (Experimental): Paclitaxel liposome injection 300mg/m2 on day 1, First cycle 28 days and subsequent cycles each 21 days
  Interventions: Drug: Paclitaxel liposome injection
- Comparator (Active Comparator): Paclitaxel injection 175mg/m2 on day 1, each 21 days
  Interventions: Drug: Paclitaxel injection

INTERVENTIONS:
Drug: Paclitaxel liposome injection
  Other Names: LIPUSU®
  Arms: Dose level A; Dose level B; Dose level C; Dose level D; Dose level E
Drug: Paclitaxel injection
  Other Names: Taxol®
  Arms: Comparator

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD)of paclitaxel liposome injection and to compare the pharmacokinetic characters between paclitaxel liposome injection and paclitaxel injection and to value the effectiveness for cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* patient willing to sign an Investigational Review Board(IRB) approved written informed consent document
* patient age: 18 years -75years
* patient must have histologically confirmed solid tumor
* patient must have uncurable and unresectable solid tumor of advanced stages
* patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* patient must have a life expectancy at least 12 weeks
* patient must have at least one lesion measurable according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.0
* patient must have progress or recurrence after at least one chemotherapy regimen for advanced stage
* patient must have adequate marrow,hepatic and renal function: defined as ANC≥2.0 × 109/L，PLT ≥10 ×109/dL, Hb ≥ 9g/dL;GOT/GPT≤2.5×ULN；Toltle bilirubin ≤1.5×ULN; Serum creatinine ≤1.5×ULN or Creatinine clearance≥40ml/min(according to Cockcroft-Gault；
* patient must have the left ventricular ejection fraction (LVEF)≥50% confirmed by ultrasonic heart scanning
* women must have the negative pregnancy test; women and men must agree to use adequate contraception

Exclusion Criteria:

* patient must non have received any other antitumor therapy, including chemotherapy, radiotherapy, hormonal therapy, biological therapy, immunotherapy and any other investigational agent within 4 weeks prior to starting study
* patient must non have any pre-existing toxity from prior antitumor therapy (any≥ grade 2, any≥1 peripheral neuropathy, excluding alopecia)
* patient must non have uncontrolled cerebral metastases
* patient must non have any uncontrolled heart illness including, but not limited to, ongoing symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, arterial hypertension (≥180/110), heart failure and myocardial infarction within 6 months prior to starting study
* Patient must not have a history of a malignancy tumor except for the following: adequately treated localized basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix for at least 5 years
* patient must non have any serious illness including, but not limited to hepatic, renal, respiratory and uncontrolled diabetes mellitus
* patient must non have psychiatric illness/social situations that would limit compliance with study requirements.
* patient must non have active or uncontrolled infection including, but not limited to tuberculosis,HIV,HBV, HCV
* Patient must non be receiving any other antitumor agent
* patient must non be pregnant and/or breastfeeding
* patient must non be receiving protease inhibitors,inhibitors of CYP3A4,antifungal agents and inducing agent of CYP3A4

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose(MTD)of paclitaxel liposome injection | completion of cycle 1(28 days)
  Graded and described using National Cancer Institute(NCI)Common Terminology Criteria for adverse events (CTCAE 4.0)

SECONDARY OUTCOMES:
dose-limiting toxicities(DLTs) of paclitaxel liposome injection | completion of cycle 1 (28 days)
  Graded and described using National Cancer Institute(NCI)Common Terminology Criteria for adverse events (CTCAE 4.0)

OTHER OUTCOMES:
Pharmacokinetic characters of paclitaxel liposome injection compared with paclitaxel injection | 0,during infusion 1.5h, 3h, after infusion 15min, 30min, 1h,2h,4h,8h,12h,24h,36h,48h,72 h
  Peak Plasma Concentration(Cmax), peak time (Tmax), Half life(T1/2), Area under the plasma concentration versus time curve(AUC0-t), Clearance (CL/F), Apparent volume of distribution(Vd/F), Mean Residence Time (MRT),

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - No.52 Fucheng Road, Haidian District,Beijing,, Beijing, Beijing Municipality